CLINICAL TRIAL: NCT05449418
Title: ENSPIRE: Engaging Staff to Improve COVID-19 Vaccination Response at Long-Term Care Facilities
Brief Title: Engaging Staff to Improve COVID-19 Vaccination Response at Long-Term Care Facilities
Acronym: ENSPIRE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Global Alliance to Prevent Prematurity and Stillbirth (GAPPS) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: R221031001
Record Dates: First submitted 2022-06-22; First posted 2022-07-08 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: COVID-19
Keywords: vaccine confidence
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Usual Care (Active Comparator): Distribution of COVID-19 vaccine promotion materials from the Centers for Disease Control and Prevention [CDC] or other national organization with limited distribution support at long-term care centers.
  Interventions: Other: Enhanced Usual Care
- Full Intervention (Experimental): Development of materials co-designed with and tailored to language/cultural affinity groups and distributed with assistance from co-design participants who will serve as peer advocates.
  Interventions: Behavioral: Full Intervention

INTERVENTIONS:
Behavioral: Full Intervention — A small group of employees who work at facilities randomized to this arm will be invited to develop tailored COVID-19 vaccination promotion materials in teams with other long-term care staff sharing the same or similar language and/or cultural affinity. These employees will also help promote these materials to all of the employees who work at their facilities.
  Other Names: Co-Design and Peer Advocacy
  Arms: Full Intervention
Other: Enhanced Usual Care — Employees who work at facilities randomized to this arm will see COVID-19 vaccine promotion materials from the Centers for Disease Control and Prevention [CDC] or other national organization.
  Arms: Enhanced Usual Care

SUMMARY:
The ENSPIRE study is a cluster-randomized comparative effectiveness trial being conducted within long-term care and residential facilities that will test a communication and engagement strategy for increasing COVID-19 booster vaccination rates against an enhanced usual care comparator (Centers for Disease Control and Prevention or other national organization vaccine education and communication materials) among facility staff. The communication and engagement strategy being tested includes (1) the development of materials co-designed with and tailored to facility staff whose primary language is a language other than English or who are from certain cultural affinity groups and (2) the distribution of the developed materials by members of the language/cultural affinity groups with peer advocacy activities (full intervention). The study is being conducted in Washington state and Georgia.

Long-term care/residential facilities will be asked to furnish their staff booster rate at 4 timepoints: pre-intervention, and one month (timepoint 1), 3 months (timepoint 2), and 6 months (timepoint 3) post-intervention. Staff at participating long-term care facilities will be invited to complete three online surveys at 3 timepoints: pre-intervention, 3 months post-intervention and 6 months post-intervention. Long-term care facilities will be randomized to a trial arm following the pre-intervention data collection.

ELIGIBILITY:
Inclusion Criteria:

* Works at a participating long-term care facility that has more than 50 staff members, has a staff COVID-19 booster vaccination rate of ≤60% as of December 1, 2021, and is located in Washington state or Georgia.
* 18 years or older

Exclusion Criteria:

* Does not work at an enrolled long-term care facility
* 17 years or younger

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 988 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in COVID-19 booster vaccination rate | Baseline (Time 0); 7 months post-randomization (Time 1); 10 months post-randomization (Time 2); 13 months post-randomization (Time 3)
  Change in percentage of staff at long-term care centers that have received a booster vaccine over time.
Change in likelihood of recommending COVID-19 vaccination | Baseline (Time 0); 10 months post-randomization (Time 2); 13 months post-randomization (Time 3)
  Change in likelihood of recommending COVID-19 vaccination to others (coworkers, family, friends) assessed using a 6-item Net Promoter Score scale. The scale is assessed on an 11-point scale ranging from 0 ('Least Likely') to 10 ('Most Likely').

SECONDARY OUTCOMES:
Change in vaccine hesitancy | Baseline (Time 0); 10 months post-randomization (Time 2); 13 months post-randomization (Time 3)
  Change in vaccine hesitancy assessed using a modified Vaccine Hesitancy Scale with 11 items. The scale is assessed on a 5-point Likert scale with answer choices ranging from 'Strongly Disagree' to 'Strongly Agree.'
Change in COVID-19 vaccine confidence | Baseline (Time 0); 10 months post-randomization (Time 2); 13 months post-randomization (Time 3)
  Change in vaccine confidence using a modified 3-item Vaccine Confidence Scale. The answer choices are on a Likert-scale: 'strongly agree', 'tend to agree', 'tend to disagree', 'strongly disagree', and 'I don't know.'

OTHER OUTCOMES:
Change in COVID-19 vaccine knowledge | Baseline (Time 0); 10 months post-randomization (Time 2); 13 months post-randomization (Time 3)
  Change in COVID-19 vaccine knowledge using 6 COVID-19 vaccine knowledge true/false questions adapted from information on the CDC's COVID-19 Myths and Facts webpage.
Change in COVID-19 vaccine attitudes | Baseline (Time 0); 10 months post-randomization (Time 2); 13 months post-randomization (Time 3)
  Change in COVID-19 vaccine attitudes using 10 questions assessed on a 5-point Likert scale adapted from existing surveys and polls assessing COVID-19 vaccine perceptions.

CONTACTS AND LOCATIONS:
Overall Officials: Clarissa Hsu, PhD, Principal Investigator — Kaiser Permanente
Locations (2):
- United States (2):
  - Kaiser Permanente Georgia Center for Research and Evaluation, Atlanta, Georgia
  - Kaiser Permanente Washington Health Research Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No